CLINICAL TRIAL: NCT06031636
Title: Observation of the Efficacy and Safety of Oncolytic Adenovirus Injection Combined With Programmed Death Receptor Inhibitors in Treatment of Advanced Malignant Pleural Mesothelioma : a Single Center, Prospective, Case Registration Study
Brief Title: Oncolytic Adenovirus(H101) Combined With PD-1 Inhibitors in Patients With Advanced Malignant Pleural Mesothelioma
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University Second Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: H101 for MPM
Record Dates: First submitted 2023-09-02; First posted 2023-09-11 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Malignant Pleural Mesothelioma, Advanced
Keywords: Malignant Pleural Mesothelioma, Advanced; Oncolytic Adenovirus; Programmed Death Receptor
MeSH Terms: conditions — Mesothelioma, Malignant

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Oncolytic adenovirus(H101) combined with PD-1 inhibitors: This study observed 2-4 treatment cycles. For the convenience of statistics, this project stipulated that the first combined medication (v1) after the patient was enrolled in this study was administered with oncolytic virus (recombinant human adenovirus type 5) by intratumoral injection or intrapleural injection on the 1-3 days. On the 4th or 5th day, PD-1 injection was administered once per cycle. The completion of two visits in this study is considered a completed case, and subsequent treatment is determined jointly by the researcher and the subject.
  Interventions: Drug: Oncolytic Adenovirus H101; Drug: Programmed death receptor-1 inhibitor

INTERVENTIONS:
Drug: Oncolytic Adenovirus H101 — The oncolytic virus(H101) is administered by intratumoral injection or intrapleural injection on days 1-3 of the first medication cycle. PD-1 inhibitor is administered on days 4 or 5, with one infusion per cycle. The treatment regimen consists of 2-4 cycles
  Other Names: Recombinant Human Type-5 Adenovirus
Drug: Programmed death receptor-1 inhibitor — The oncolytic virus(H101) is administered by intratumoral injection or intrapleural injection on days 1-3 of the first medication cycle. PD-1 inhibitor is administered on days 4 or 5, with one infusion per cycle. The treatment regimen consists of 2-4 cycles

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Oncolytic Adenovirus(H101) combined with PD-1 inhibitor in patients with advanced malignant pleural mesothelioma who have previously been resistant to advanced PD-1 inhibitors.

DETAILED DESCRIPTION:
By monitoring the clinical symptoms of patients with advanced immune resistant pleural mesothelioma treated with adenovirus injection combined with programmed death receptor (PD-1) inhibitors, we analyze and explore the effectiveness and safety of using oncolytic virus drugs. Exploring the influencing factors of using oncolytic adenovirus injection combined with PD-1 inhibitors to reverse immune resistance in MPM patients. Evaluate the safety of the drug, and finally evaluate the quality of life of patients using oncolytic adenovirus injection(H101) combined with PD-1 inhibitors.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old (including boundary values), regardless of gender.
2. Confirmed as late stage MPM patients who have failed immunotherapy.
3. The patient or their legal representative can understand and sign the informed consent form.
4. At least one lesion that can safely undergo intratumoral injection or intrapleural injection of oncolytic adenovirus as the target lesion, with a diameter of spiral CT ≥ 1cm or ordinary CT ≥ 2cm, and can be measured through imaging methods.
5. ECOG score 0-2.

Exclusion Criteria:

1. Physicians participating in the study believe that patients may not be able to provide continuous follow-up information.
2. Any uncontrollable clinical problems (such as severe mental, neurological, cardiovascular, respiratory, and other systemic diseases).
3. Contraindications to relevant drugs (such as oncolytic adenoviruses, PD-1 inhibitors, etc.)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with malignantpleural mesothelioma who have previously been resistant to advanced PD-1 inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-07-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
ORR(Objective Response Rate) | 36 months
  The proportion of CR(complete response) and PR(partial response) in all patients.
DCR(Disease Control Rate) | 36 months
  The proportion of CR(complete response), PR(partial response) and SD(stable disease) in all patients.

SECONDARY OUTCOMES:
PFS(Progression Free Survival) | 36 months
  Refers to the time from the first treatment day to the first occurrence of disease progression or death from any cause (whichever occurs first), and the end point event is determined by the investigator according to RECIST version1.1.
OS(Overall Survival) | 36 months
  Time between the date of grouping and death from any cause or the end of the last follow-up visit.
AEs(Adverse Events) | 36 months
  Toxicity were graded according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE), version 5.0. All serious and non-serious adverse events that occur after enrollment through 30 (+7) days after the last administration of H101 will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical Unversity Second Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided